CLINICAL TRIAL: NCT03912038
Title: Non-caloric Sweeteners Levels in Breast Milk and Newborn's Blood and Effect on Microbiota's Composition.
Status: Completed | Type: Observational
Sponsor: Hospital General de México Dr. Eduardo Liceaga (Other Government)
Responsible Party: Principal Investigator, Marcela Esquivel V, Medical Sciences Researcher, Hospital General de México Dr. Eduardo Liceaga
Other Study IDs: DI/17/301/05/075
Record Dates: First submitted 2019-04-08; First posted 2019-04-11 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Microbial Colonization
Keywords: Non-caloric sweeteners; microbiota; breast milk; umbilical cord
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma Feces Breast milk Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Null or low consumption: No-intervention. The group consists of women who have reported a null or low consumption of non-caloric sweeteners during late pregnancy.
  Interventions: Other: No intervention.
- Moderate consumption: No-intervention. The group consists of women who have reported a moderate consumption of non-caloric sweeteners during late pregnancy.
  Interventions: Other: No intervention.
- High consumption: No-intervention. The group consists of women who have reported a high consumption of non-caloric sweeteners during late pregnancy.
  Interventions: Other: No intervention.

INTERVENTIONS:
Other: No intervention. — No intervention

SUMMARY:
This study evaluates the presence and quantity of non-caloric sweeteners in newborns umbilical cord blood, and in their mother's breast milk at delivery, at 2 months, 4 months and 6 months of age. Microbiota composition will be evaluated in milk and in feces of both mother and child.

DETAILED DESCRIPTION:
The consumption of non-caloric sweeteners (ENC) is increasingly common in our country due to its wide use in all types of food and beverages, even those not labeled as "diet". Despite its widespread use and being an alternative to the consumption of sugars, several studies have shown that frequent ENC users are also at risk of excessive weight gain, type II diabetes, and cardiovascular diseases. In addition to this, the consumption of ENC in the early stages of life may predispose to the development of metabolic disorders later in life.The ENC have been shown to have effects on the health of those who consume them, causing metabolic disorders, weight gain and changes in the microbiota. The newborns, in whom gut microbiota is in the process of being established, influenced by the vaginal and intestinal microbiota of the mother, as well as by the mother's milk, are a vulnerable population in whom the effect of ENC consumption has not been investigated. This makes it relevant to study the prevalence of ENC in breast milk and umbilical cord blood of their newborns and to evaluate the composition of the intestinal and milk microbiota in order to identify changes attributable to the consumption of ENC.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40 years old
* Women in labor
* Consent to participate in the study

Exclusion Criteria:

* Pre-term delivery (<30 weeks)
* Metabolic diseases (insulin resistance, diabetes, gestational diabetes)
* Hypertension
* Thyroid disease
* Cancer

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women in labor who come to the service of gynecology and obstetrics General Hospital Mexico. Usually, they are residents from Mexico City and metropolitan area (Mexico State).
Sampling Method: Non-Probability Sample
Enrollment: 178 (Actual)
Dates: Start 2018-01-26 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Microbiota composition in feces | 2 months
  Composition of feces microbiota in mother and newborn
Microbiota composition in feces | 4 months
  Composition of feces microbiota in mother and newborn
Microbiota composition in feces | 6 months
  Composition of feces microbiota in mother and newborn
Microbiota composition in breast milk | 0 months
  Composition of breast milk microbiota
Microbiota composition in breast milk | 2 months
  Composition of breast milk microbiota
Microbiota composition in breast milk | 4 months
  Composition of breast milk microbiota
Microbiota composition in breast milk | 6 months
  Composition of breast milk microbiota
Non-caloric sweeteners levels at birth | at birth
  Non-caloric sweeteners levels in milk, plasma, umbilical cord plasma, urine in mg/mL
Non-caloric sweeteners levels 2 months follow-up | 2 months after birth
  Non-caloric sweeteners levels in breast milk and urine in the 2 months follow-up
Non-caloric sweeteners levels 4 months follow-up | 4 months after birth
  Non-caloric sweeteners levels in breast milk and urine in the 4 months follow-up
Non-caloric sweeteners levels 6 months follow-up | 6 months after birth
  Non-caloric sweeteners levels in breast milk and urine in the 6 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Marcela Esquivel, PhD, Principal Investigator — Hospital General de México Dr. Eduardo Liceaga
Locations (1):
- General Hospital of Mexico Dr. Eduardo Liceaga, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided